CLINICAL TRIAL: NCT07106697
Title: Video-Assisted First Aid by Young Children for Unconsciousness
Brief Title: Video-assisted First Aid by Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Video-assisted first aid
Record Dates: First submitted 2025-07-21; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Unconsciousness
Keywords: unconsciousness; dispatcher-assistance; children; video-guidance
MeSH Terms: conditions — Unconsciousness

STUDY DESIGN:
Intervention Model Description: Children were allocated in pairs to one of three parallel intervention arms:
  Training combined with video-guided assistance,
  Video-guided assistance only, or
  No intervention (control). Each pair participated in only one intervention condition without crossover. Parallel assignment allowed for comparison of outcomes between intervention strategies and the control group. Video guidance was provided live by a trained dispatcher during simulation scenarios.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The dispatcher, assessors, actor, and children were informed about their specific tasks according to their group allocation but were blinded to the study design and intended outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Training and video-assistance (Experimental): Received a 45-minute theoretical and practical training session on assessing unconsciousness and managing an unresponsive victim, based on ILCOR first aid guidelines, followed by a 15-minute technical session on how to initiate and operate video assistance via a smartphone. Both sessions were conducted by a paramedic experienced in pediatric first aid education and emergency dispatching.
  Interventions: Behavioral: First Aid Training Combined With Video-Assisted Guidance
- Video-assistance only (Experimental): Received a 15-minute technical session exclusively focused on operating the video assistance technology (without first aid instruction). This session was conducted by the same paramedic as in Group 1.
  Interventions: Behavioral: Video-Assisted Guidance Without Prior Training
- No assistance (No Intervention): Received no preparatory training (control group).

INTERVENTIONS:
Behavioral: First Aid Training Combined With Video-Assisted Guidance — Participants received a 45-minute structured first aid training session on unconscious victim management, followed by a 15-minute video-guidance instruction. During simulation, children received real-time video guidance from a dispatcher via smartphone.
  Arms: Training and video-assistance
Behavioral: Video-Assisted Guidance Without Prior Training — Participants received a 15-minute instruction on video-assisted guidance use, without prior first aid training. During simulation, real-time video guidance was provided by a dispatcher via smartphone to assist with first aid tasks.
  Arms: Video-assistance only

SUMMARY:
Sudden cardiac arrest is a major public health issue, and EMS dispatchers play a key role in improving outcomes through telephone-assisted CPR (T-CPR). With current technology, video-assisted CPR (V-CPR) via smartphones allows for visual feedback and more precise guidance. While V-CPR has shown promise, studies have mostly focused on adult CPR performance in controlled settings. Research involving children and non-CPR first aid scenarios is scarce. Our study addresses this gap by evaluating video-assisted guidance during a simulated unconsciousness situation performed by children, exploring its feasibility and broader applicability.

DETAILED DESCRIPTION:
Sudden cardiac arrest is a major public health concern and remains one of the leading causes of death in industrialized countries. Emergency Medical Services (EMS) dispatchers play a crucial role in recognizing cardiac arrest and guiding lay responders through telephone-assisted CPR (T-CPR), which has been shown to improve survival outcomes. With current technologies, real-time video communication via a bystander's smartphone has become feasible, enabling video-assisted CPR (V-CPR), which allows dispatchers to provide visual feedback and more tailored guidance.

Although several studies have investigated the effectiveness of V-CPR-mainly in terms of chest compression quality and time to first compression-these have primarily focused on adult participants and controlled settings. Research involving children as lay responders is limited, and video-assisted first aid has been scarcely evaluated in pediatric populations. Moreover, existing studies concentrate predominantly on CPR, while other essential first aid scenarios, such as the management of unconscious victims, remain underexplored.

To address these gaps, our study examined the effectiveness of video-assisted guidance during a simulated unconsciousness scenario performed by children, aiming to assess both the feasibility and potential benefits of extending video-assisted firs aid approaches beyond cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* healthy children aged 6 to 8 years (first grade of primary school)

Exclusion Criteria:

* children with known physical, cognitive, or communication impairments that could interfere with participation in simulated first aid tasks
* technical issue during data collection

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Correctness of treatment of an unconscious patient (based on a checklist). | During post-analysis of the video-records (within 1 week after data collection)
  Number of correct first aid steps performed and task completion success (based on the checklist containing all the relevant steps of the treatment).

SECONDARY OUTCOMES:
Time | During procedure.
  Time to task completion

OTHER OUTCOMES:
Helping attitude of the children (based on willingness to help). | During procedure.
  Observable willingness to help (approach and engagement behavior during the simulated procedure). The proportion of children who dared to approach the victim and initiate care in the simulated scenario was measured. Based on this, participants were classified into "positive" and "negative" attitude groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pécs Faculty of Health Sciences, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No